CLINICAL TRIAL: NCT06709911
Title: Efficacy of Multimodal Interventions for Tenosynovitis: Comparative Analysis of Basic Manipulation, Tui Na, Blood Flow Restriction Training, and Magnetic Bead Application Combined With Tui Na
Brief Title: A Comparative Study of the Efficacy of Multimodal Interventions for Tenosynovitis
Acronym: TGCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zixin Deng (Other)
Responsible Party: Sponsor-Investigator, Zixin Deng, Sponsor-Investigator, First People's Hospital of Foshan
Organization: First People's Hospital of Foshan (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: University of Leeds
Record Dates: First submitted 2024-11-17; First posted 2024-11-29 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: TGCT
MeSH Terms: interventions — Massage; Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Basic Manipulation Stretching Group (Experimental): Focuses on relieving muscle tension and tendon adhesions in the flexor and extensor muscles of the wrist and hand. The intervention aims to improve soft tissue elasticity, enhance joint mobility, and restore functional wrist and hand movement through systematic stretching techniques.
  Interventions: Behavioral: Basic Manipulation Stretching
- Massage and Tui Na Manipulation (Experimental): Uses a combination of massage and Tui Na techniques to target tendon sheaths and surrounding tissues in the wrist and hand. Specific acupoints, such as Hegu, Yangchi, and Waiguan, are stimulated to alleviate inflammation, improve blood circulation, and restore joint functionality. The intervention aims to enhance soft tissue elasticity and range of motion while reducing pain and stiffness.
  Interventions: Behavioral: Massage and Tui Na Manipulation
- Blood flow restriction training group (Experimental): Applies localized blood flow restriction using pressurized equipment on the proximal forearm, combined with low-load exercises such as wrist flexion, extension, clenching, and rotation. The goal is to stimulate muscle adaptation and strength development while minimizing mechanical stress on the joints, ultimately improving hand and wrist functionality.
  Interventions: Behavioral: Blood flow restriction training
- Magnetic Bead Pressure Stimulation and Tui Na Manipulation Combined Intervention Group (Experimental): Combines magnetic bead pressure stimulation and Tui Na manipulation to enhance therapeutic outcomes. Magnetic beads are applied to specific acupoints on the hand and wrist (e.g., Hegu, Ashi, Waiguan) to stimulate circulation and reduce tension. Tui Na techniques, including pressing, kneading, and massaging, further enhance the stimulation, alleviate inflammation, reduce tendon adhesions, and promote mobility recovery.
  Interventions: Behavioral: Magnetic Bead Pressure Stimulation and Tui Na Manipulation Combined Intervention

INTERVENTIONS:
Behavioral: Basic Manipulation Stretching — This group received standard hand tenosynovitis stretching therapy, which focused on the flexor and extensor muscle groups of the wrist and hand for release. Muscle tension and tendon adhesions were relieved by basic stretching maneuvers, with each intervention lasting 20-30 minutes, twice a week, over a 4- to 8-week period.
  Arms: Basic Manipulation Stretching Group
Behavioral: Massage and Tui Na Manipulation — The group received Tui Na manipulation interventions, including pointing, pressing and rolling techniques for the tendon sheath and thumb region, focusing on the stimulation of acupoints such as Hegu, Yangchi and Waiguan. The aim of Tui Na manipulation was to relieve the inflammatory reaction around the tendon sheath, promote blood circulation and improve local function. Each intervention lasts 20-30 minutes, twice a week for 4-8 weeks.
  Arms: Massage and Tui Na Manipulation
Behavioral: Blood flow restriction training — This group used pressurized blood flow restriction training, in which the proximal part of the temporal joint was pressurized by a pressurized device to restrict blood flow. The training consisted of low-load wrist flexion and extension, fist clenching and unclenching, and wrist rotation. The training intensity was set at 20%-50% 1RM, and the frequency was 2 times per week for 4 to 8 weeks. Pressurization was performed before training and the pressure was set in the range of 20-50 mmHg, and the training period was supervised by a professional.
  Arms: Blood flow restriction training group
Behavioral: Magnetic Bead Pressure Stimulation and Tui Na Manipulation Combined Intervention — This group received the combined intervention of magnetic bead pressure stimulation and Tui Na manipulation. Before treatment, the magnetic beads were applied to specific acupoints on the hand (e.g., Hegu, Ahshi, Waiguan, etc.), fixed by breathable patches, and combined with Tui Na manipulation. During Tui Na, the magnetic beads are pressed and kneaded to further enhance the stimulation effect of the acupoints. After Tui Na, the magnetic beads remain in the affected area and can be pressed and kneaded 2-3 times a day for 3 minutes each time to produce a slight sensation of soreness and distension. The aim of the massage is to relieve the inflammatory reaction around the tendon, loosen muscle tension and tendon sheath adhesions and promote blood circulation and joint mobility. The cycle of intervention is 4 to 8 weeks.
  Arms: Magnetic Bead Pressure Stimulation and Tui Na Manipulation Combined Intervention Group

SUMMARY:
The goal of this clinical trial is to compare the efficacy of four treatments in patients with hand tenosynovitis. The main questions it aims to answer are:

Which treatment most effectively reduces pain and improves joint function? How do the treatments differ in improving strength and range of motion? Researchers will compare four groups-basic manipulation, tui na manipulation, blood flow restriction (BFR) training, and magnetic bead application combined with tui na-to see if there are differences in clinical outcomes.

Participants will:

Be randomly assigned to one of the four treatment groups. Receive interventions twice a week for 4-8 weeks. Undergo assessments of pain, function, range of motion, and strength before, during, and after the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age.
* Case diagnosis reporting symptoms of tenosynovitis of the hand for at least 3 months.
* Constant-Murley Shoulder Score: score less than or equal to 60.
* Dysfunction of the Upper Extremity, Shoulder, and Hand Scale (DASH Scale): DASH score less than 40.
* Mayo Wrist Score: score less than or equal to 60.
* Positive test results on 2 or more scales during pre-test screening.
* No structural lesions or congenital malformations of the hand or wrist.
* Finkelstein's Test: Positive (pain occurs when patient holds thumb and bends wrist toward little finger).
* Fist Clenching Test: Positive (pain increases when patient clenches fist and attempts to bend wrist toward little finger).
* No prior hand or wrist surgery or external injuries.
* No serious cardiac, pulmonary, neurological, or other systemic diseases.
* Sufficient exercise capacity to complete exercise loads of required intensity and duration.

Exclusion Criteria:

* Not between 18 and 60 years of age.
* Failed wrist function screening.
* Failed special tests.
* Presence of structural wrist lesions or congenital wrist deformities.
* History of wrist surgery, significant trauma, or wounds.
* Problems with skin irritation, infections, or open wounds.
* Conditions like anemia or low blood pressure.
* Serious cardiac, pulmonary, neurological, or other systemic diseases.
* Inability to cooperate with trial requirements or refusal to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale, VAS | Baseline, 4 weeks (after Week 4 of treatment), 8 weeks (after the final treatment at Week 8)
  The VAS score consists of five dimensions of pain threshold testing: overall wrist pain, pain when extending the wrist, pain when flexing the wrist, wrist pain when resisting forearm rotation, and pain when pressing on specific parts of the wrist. Each dimension is scored on a scale of 0-10 for a total of 50 points, with lower scores indicating less pain.
Mayo Wrist Score, MWS | Baseline, 4 weeks (after Week 4 of treatment), 8 weeks (after the final treatment at Week 8)
  The scale consists of four areas: pain (25 points), function (25 points), range of motion (25 points), and grip strength (25 points) for a total of 100 points, with higher scores indicating better wrist function.
Wrist strength | Baseline, 4 weeks (after Week 4 of treatment), 8 weeks (after the final treatment at Week 8)
  An electronic grip strength device was used to measure the grip strength of the affected arm before and after the treatment, including the grip strength of the affected arm in three states; the maximum grip strength in the naturally hanging arm state, the maximum grip strength in resisted internal rotation of the forearm, and the maximum grip strength in resisted external rotation of the forearm.
Range of Motion Measurement | Baseline, 4 weeks, (after Week 4 of treatment), 8 weeks (after the final treatment at Week 8)
  Flexion and extension angle measurements, forearm pronation and pronation angle measurements

CONTACTS AND LOCATIONS:
Overall Officials: Xin Z Deng, Principal Investigator

IPD SHARING:
Plan to Share IPD: No